CLINICAL TRIAL: NCT05966064
Title: DEnosumab for the Treatment of FIbrous Dysplasia/McCune-Albright Syndrome in Adults (DeFiD): a Randomized Double-blind Placebo-controlled Trial
Brief Title: DEnosumab for the Treatment of FIbrous Dysplasia/McCune-Albright Syndrome in Adults (DeFiD)
Acronym: DeFiD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Natasha Appelman-Dijkstra (Other)
Responsible Party: Sponsor-Investigator, Natasha Appelman-Dijkstra, Principal investigator, Internist-Endocrinologist, MD, PhD, Leiden University Medical Center
Organization: Leiden University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022-501705-12-00
Record Dates: First submitted 2023-06-19; First posted 2023-07-28 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Fibrous Dysplasia; McCune Albright Syndrome
MeSH Terms: conditions — Fibrous Dysplasia of Bone; Fibrous Dysplasia, Polyostotic | interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Denosumab (Active Comparator): Denosumab randomized at baseline and 3 months in a double-blinded fashion and in case of open label at 6 and 9 months
  Interventions: Drug: Denosumab 120 Mg/1.7 Ml Inj
- Placebo (Placebo Comparator): Placebo randomized at baseline and 3 months in a double-blinded fashion.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Denosumab 120 Mg/1.7 Ml Inj — Denosumab randomized at baseline and after 3 months at 6 and 9 months in case of open label
  Other Names: Xgeva
  Arms: Denosumab
Drug: Placebo — placebo randomized at baseline and after 3 months
  Arms: Placebo

SUMMARY:
Fibrous Dysplasia/McCune-Albright syndrome (FD/MAS) is a rare disease, consisting of the replacement of normal bone tissue with fibrous tissue. FD lesions may be isolated in one or more bones or may be associated with endocrinopathies in McCune-Albright syndrome. Bone lesions constitute of weak bone tissue, leading to higher risk of fractures, pain and decreased quality of life. There is no cure for FD lesions and current therapies failed to soothe patients' complaints or to display any effect on progression of the lesions on imaging. However, the RANKL-inhibitor Denosumab demonstrated encouraging results in mouse models and in off-label clinical use, leading to clinical, biochemical and radiographical improvements.

Study's aim is to investigate whether 3-monthly Denosumab will improve the clinical, radiological and biochemical manifestations of FD bone lesions.

DETAILED DESCRIPTION:
Eligible patients will be randomized to treatment with either subcutaneous Dmab 120mg or placebo at baseline and 3 months in a blinded fashion. At 6 months, after 2 injections, patients with pain score <4 will exit the study to discontinue study medication and proceed in usual care, while patients with pain score ≥4 or lesional growth will be offered Dmab 120 mg at 6 and 9 months in an open-label design.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic patients with established diagnosis of FD/MAS and closed growth plates(>18 years)
* Pain in the region of an FD localization, not responding to adequate pain treatment and without mechanical component e.g. impending fracture
* Pain score from FD lesion for maximum or average pain on VAS ≥ 4
* Increased lesional activity defined as increased bone turnover markers (ALP, P1NP or CTX) or increased activity on Na[18F]-PET/CT or bone scintigraphy in at least one lesion
* Normal levels of calcium, parathyroid hormone and vitamin D (supplementation is allowed)
* Treated hypophosphatemia (defined as >0.7 at two separate measures)
* good dental health (last check within the last 12 months)

Exclusion Criteria:

* Active pregnancy wish, pregnancy or nursing
* Pain not related to FD
* Uncontrolled endocrine disease
* Untreated vitamin D deficiency, hypocalcemia or hypophosphatemia
* Previous use of bisphosphonates or Dmab < 6 months before inclusion ('6 months wash out')
* Previously reported severe side effects on Dmab
* Inability to fulfil study requirements
* Poor untreated dental health without intention to get treatment
* Treatment with other bone influencing drugs, such as high doses corticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2023-06-13 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Denosumab effect on maximal pain score | at baseline, 3 months and after 6 months and in case of open label treatment after 9 and 12 months
  Evaluation of maximal pain score changes after treatment, assessed by Brief Pain Inventory (scale 0 to 10; 0-no pain, 10 worst pain)

SECONDARY OUTCOMES:
Denosumab effect on average pain scores | at baseline, 3 months and after 6 months and in case of open label treatment after 9 and 12 months
  Evaluation of average pain score changes after treatment, assessed by Brief Pain Inventory (scale 0 to 10; 0-no pain,10 worst pain)
To evaluate the number of patients with 50% reduction of maximal pain (BPI) | at baseline, 3 months and after 6 months and in case of open label treatment after 9 and 12 months
  Evaluation of the number of patients with 50% reduction of maximal pain score changes after treatment, asseses by Brief Pain Inventory (scale 0 to 10; 0-no pain, 10 worst pain)
Denosumab effect on quality of life | at baseline, 3 months and after 6 months and in case of open label treatment after 9 and 12 months
  Evaluation of Denosumab effect on quality of life, assessed with validated questionnaire SF-36 (scale 0-100, higher scores indicate better health status)
Denosumab effect on average weekly pain score | every week from baseline, through study completion, an average of 1 year
  Evaluation of Denosumab effect on average weekly pain score assessed through a pain diary with VAS score (scale 0 to 10)
Denosumab effect on Physical activity assessment assessed through Health Assessment Questionnaire - Disability Index | baseline, 3 months and 6 months, and in case of open label treatment after 9 and 12 months
  Evaluation of Denosumab effect on on Physical activity assessment (Health Assessment Questionnaire - Disability Index: Health state index scores generally range from less than 0 (where 0 is a health state equivalent to death; negative values are valued as worse than death) to 1 (perfect health), with higher scores indicating higher health utility, though health state preferences can differ between countries.
Denosumab effect on Physical activity assessment assessed through screenshot of pedometer | baseline, 3 months and 6 months, and in case of open label treatment after 9 and 12 months
  Evaluation of Denosumab effect on on Physical activity assessment ( screenshot of pedometer of activity during the last week on smartphone, unit measure: number of steps during the last week)
Evaluation of prevalence of possible neuropathic component of the reported pain | baseline, 3 months and 6 months and in case of open label treatment after 9 and 12 months
  to evaluate the prevalence of possible neuropathic component of the reported pain through Pain Detect questionnaire (It is scored from 0 to 38, with total scores of less than 12 considered to represent nociceptive pain, 13-18 possible NeP, and >19 representing >90% likelihood of Neuropathic pain)
To investigate the number of analgesics used for pain | baseline, 3 months and 6 months and in case of open label treatment after 9 and 12 months
  number of used analgesics for pain : unit of measure: number
To investigate the frequency use of analgesics for pain | baseline, 3 months and 6 months and in case of open label treatment after 9 and 12 months
  the frequency use of analgesics for pain (daily, multiple times per day, multiple times per week, monthly, when necessary)
To investigate the dosage of analgesics used for pain | baseline, 3 months and 6 months and in case of open label treatment after 9 and 12 months
  dosage of analgesics used for pain (unit of measure: mg)
Denosumab effect on serum bone markers | baseline, 3 months and 6 months and in case of open label treatment after 9 and 12 months
  effect of denosumab on bone serum markers (alkaline phosphatase (measure unit: U/L), P1NP -Procollagen-1-propeptide (measure unit: ng/ml), Beta-crosslaps (measure unit: ug/L)
Denosumab effect on serum markers | baseline, 3 months and 6 months and in case of open label treatment after 9 and 12 months
  effect of Denosumab on serum calcium(mmol/L), fosfate (mmol/L), PTH (pmol/L)
Denosumab effect on lesion size | baseline and after 6 months, and in the case of open label treatment after 12 months
  Na18F-PET/CT scan- measurement of lesion size
Denosumab effect on lesion activity | baseline and after 6 months, and in the case of open label treatment after 12 months
  Na18F-PET/CT scan- ,measurement of Na18F uptake
disease quantification (Skeletal Burden Score (SBS) | at baseline, 6 months and after 12 months
  nuclear imaging ((Skeletal Burden Score (SBS): scale 0 to 75, higher scores meaning increased disease activity
Denosumab effect on bone density | baseline and after 12 months
  Dual-energy X-ray absorptiometry (DXA) - bone density measurement ( T-score of -1.0 or above = normal bone density T-score between -1.0 and -2.5 = low bone density, or osteopenia; T-score of -2.5 or lower = osteoporosis)
Denosumab effect on vertebral fractures | baseline and after 12 months
  Dual-energy X-ray absorptiometry (DXA) - assement of presence of Vertebral Fractures through Vertebral Fractures Assessment (VFA) and changes from baseline until 12 months after
To assess potential side effects in the form of Atypical femoral fractures | after 12 months
  Dual-energy X-ray absorptiometry (DXA) femur extended

CONTACTS AND LOCATIONS:
Overall Officials: Natasha Appelman-Dijsktra, MD, PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands